CLINICAL TRIAL: NCT02205099
Title: A Single-center, Randomized, Double-blind, Flexible-dosage, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of Multiple Oral Doses of SKL15508 in Subjects With Stable Schizophrenia
Brief Title: A Safety, Tolerability, PK and PD Study of Multiple Oral Doses of SKL15508 in Subjects With Stable Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SKL15508C003
Record Dates: First submitted 2014-07-22; First posted 2014-07-31 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SKL15508 High Dose (Experimental): SKL15508 High Dose
  Interventions: Drug: SKL15508
- SKL15508 Medium Dose (Experimental): SKL15508 Medium Dose
  Interventions: Drug: SKL15508
- SKL15508 Low Dose (Experimental): SKL15508 Low Dose
  Interventions: Drug: SKL15508
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SKL15508
  Arms: SKL15508 High Dose; SKL15508 Low Dose; SKL15508 Medium Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a single-site, randomized, double-blind, placebo-controlled, multiple dose, flexible dosage range, PK and PD study of SKL15508 as monotherapy in subjects with stable schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or, when applicable, the subject's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
2. Participants who are nonsterile and sexually active agree to use a double-barrier method of contraception (must be used regardless of any other contraception in use) from the time of providing informed consent throughout the duration of the study and for 12 weeks after the last dose of study drug. Nonsterile males must be advised not to donate sperm and women should not donate ova throughout the duration of the study and for 12 weeks after the last dose of study drug.
3. Must be male or non-pregnant, non-lactating female subjects, 18 to 60 years of age, inclusive
4. Has a body mass index (BMI) between 18.0 and 38.0 kg/m2, inclusive
5. Has a clinical diagnosis of schizophrenia and, in the opinion of the Investigator, is able to safely be off his or her prescribed antipsychotic medications while participating in the study and has a very high likelihood of not deteriorating over a 3-week timeframe when off standard of care as outpatients during the Screening Period
6. Has been receiving a stable dose of antipsychotic medication for at least 1 month before Screening
7. Has not had an acute exacerbation of psychosis or hospitalization for the treatment of schizophrenia for at least 3 months before Screening
8. By history, has not had a marked change in smoking or tobacco/nicotine use from 30 days before Screening.
9. Must reside in a stable residence for at least 8 weeks before the Screening Visit

Exclusion Criteria:

1. At risk of suicide (e.g., per Columbia Suicide Severity Rating Scale [C-SSRS]) or have made a suicide attempt in the 6 months before Screening
2. Has a known sensitivity to sulfur-containing drugs or sulfates in food
3. Taking any medication known to influence coagulation, such as acetylsalicylic acid (aspirin), and including prescription, herbal remedies, vitamin supplements and over-the-counter products
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal or endocrine disease or other abnormality (other than the disease being studied), which may impact the ability of the subject to participate or potentially confound the study results
5. Has a positive urine drug result for drugs of abuse (i.e., illicit, illegal or without valid prescription or medical need) at Screening or Admission
6. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 45 days before Day 1
7. Has an abnormal (clinically significant) electrocardiogram (ECG) at Screening or unit admission day
8. Has a blood pressure and pulse rate outside the protocol defined ranges
9. Has a QT interval or PR outside of the protocol defined ranges
10. Has abnormal laboratory values that suggest a clinically significant underlying disease
11. Has a history of a primary DSM-IV axis I diagnosis other than schizophrenia
12. Has a medical condition other than schizophrenia (e.g., dementia, antisocial personality, borderline personality disorders) that can cause cognitive impairment or interfere with the performance or completion of study-defined procedures
13. Has been taking medication for a medical condition for less than 2 months even if at a stable dose or regimen
14. Currently taking lithium or any psychotropic medication that cannot be discontinued for safety reasons

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number and percent of subjects experiencing an adverse event. | 10 days
Change from baseline in event-related potentials (ERP) following multiple oral doses of SKL15508. | During the course of 10 days
Change from baseline in clinical laboratory assessments. | 10 days
Change from baseline in vital signs. | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Glendale Adventist Medical Center, Glendale, California, United States